CLINICAL TRIAL: NCT02655497
Title: Maintaining Independence in Everyday Life Among Seniors With Subjective Cognitive Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Deirdre Dawson, Senior Scientist, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB#15-29
Record Dates: First submitted 2015-11-17; First posted 2016-01-14 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Aging
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Training (Experimental): Cognitive training intervention. The intervention includes seven 2-hour group sessions interspersed with four individual 45-minute sessions for a total of 17 hours of intervention over an 8-week period. The experimental group will receive real-world strategy training, a cognitive strategy based approach that trains people to improve their level of independence on meaningful activities of daily life with which they are having difficulty.
  Interventions: Behavioral: Cognitive training
- Psychosocial education (Active Comparator): The intervention includes seven 2-hour group sessions interspersed with four individual 45-minute sessions for a total of 17 hours of intervention over an 8-week period. The control group will receive brain-health education.
  Interventions: Behavioral: Psychosocial education

INTERVENTIONS:
Behavioral: Cognitive training
  Arms: Cognitive Training
Behavioral: Psychosocial education
  Arms: Psychosocial education

SUMMARY:
The purpose of this study is to determine the effectiveness of cognitive strategies in improving participation in daily activities within older adults who report subjective cognitive decline.

DETAILED DESCRIPTION:
The planned project explores the effects of several interventions designed to promote independence in everyday life, with older adults who identify cognitive complaints. Evidence suggests that 25-50% of community dwelling older adults report cognitive difficulties, such as reduced memory or concentration, in the absence of any diagnosed condition. Cognitive skills are crucial to living independently. The investigators plan to examine two approaches in a randomized controlled trial. Based on our successful pilot study, the investigators hypothesize that this training which combines education on healthy lifestyles and problem solving training to address everyday life difficulties, will be effective in maximizing and maintaining independence of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults aged 60+
* Fluent in written and spoken English
* Have subjective cognitive complaints (SCC)
* Performance within normal limits on a neuropsychological assessment battery
* Participants must also be able to self-identify specific areas of difficulty in their everyday life that they would like to improve

Exclusion Criteria:

* Significant neurological or psychiatric history (e.g., multiple sclerosis, psychiatric illness requiring hospitalization)
* Concurrent depression
* Anaesthesia in previous 6 months; and substance abuse

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in the Canadian Occupational Performance Measure (COPM) scores | 8 weeks after pretest and 3 months after intervention finished
  The Canadian Occupational Performance Measure (COPM) is the primary outcome measure. All participants will identify five everyday life activities that they need to or want to do using the COPM. The primary outcome will be (a) the number of goals improved by two points.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Dawson, PhD, Principal Investigator — Baycrest Health Sciences
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada